CLINICAL TRIAL: NCT02225210
Title: Effects of Dexmedetomidine Sedation on Delirium and Haemodynamic in Mechanical Ventilated Elderly Patients -a Single Center,Randomized and Controlled Trial
Brief Title: Effects of Dexmedetomidine Sedation on Delirium and Haemodynamic in Mechanical Ventilated Elderly Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fuling Central Hospital of Chongqing City (Other)
Responsible Party: Principal Investigator, Shuaiya, physician, Fuling Central Hospital of Chongqing City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shu 2014
Record Dates: First submitted 2014-08-22; First posted 2014-08-26 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Safety of Dexmedetomidine Sedation
Keywords: Dexmedetomidine ,Delirium ,Haemodynamic, Mechanical ventilation
MeSH Terms: interventions — Dexmedetomidine; Midazolam; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group dexmedetomidine ,dexmedetomidine (Experimental): Continuous pump infusion dexmedetomidine with loading dose of 0.4μg.kg-1 for 10 minutes ,then followed by maintenance dose of 0.2~0.7µg.kg-1 to maintain Sedation-Agitation Scale between 3 and 4.
  Interventions: Drug: Dexmedetomidine
- Group midazolam,midazolam,fentanyl (Active Comparator): Quickly inject midazolam and fentanyl with loading dose of 0.1mg.kg-1 and 1 μg.kg-1 separately until attaining Sedation-Agitation Scale between 3 and 4,then followed by maintenance dose of 0.05~0.1mg.kg-1.h-1 and fentanyl 0.5~1μg.kg-1.h-1 separately.
  Interventions: Drug: Midazolam; Drug: Fentanyl

INTERVENTIONS:
Drug: Dexmedetomidine — Loading dose:0.4μg.kg-1 Maintenance dose :0.2~0.7µg.kg-1 Sedation-Agitation Scale: maintain between 3 and 4.
  Arms: Group dexmedetomidine ,dexmedetomidine
Drug: Midazolam — Loading dose of midazolam:0.1mg.kg-1 . Maintenance dose of midazolam :0.05~0.1mg.kg-1.h-1 . Sedation-Agitation Scale: maintain between 3 and 4
  Arms: Group midazolam,midazolam,fentanyl
Drug: Fentanyl — Loading dose of fentanyl:1 μg.kg-1 . Maintenance dose of fentanyl: 0.5~1μg.kg-1.h-1 . Sedation-Agitation Scale: maintain between 3 and 4
  Arms: Group midazolam,midazolam,fentanyl

SUMMARY:
This study was designed to observe the effects of dexmedetomidine on delirium and haemodynamic in mechanical ventilated elderly patients,and to evaluate the safety of dexmedetomidine.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Intensive care unit patients who need mechanical ventilation
* Anticipate duration of mechanical ventilation longer than 24 hours,and shorter than 96 hours prior to giving investigational products
* Acute physiology and chronic health evaluation II score more than 10
* Aged between 60 to 80 years old
* Weight between plus or minus 20% of the standard weight. Male: (height cm - 80) × 70% = standard weight Female: (height cm - 70) × 60% = standard weight

Exclusion Criteria:

* Trauma and burn patients
* Any kind of dialysis
* Suspected or confirmed difficult airway
* Use of neuromuscular blocking drugs(Except using for intubation )
* Neuromuscular disease
* Epidural or subarachnoid anesthesia
* Plan to give general anesthesia before 24 hours drugs intervention or after giving investigational drugs
* Serious central nervous system disease
* Mental disability or mental disease
* Acute hepatitis and serious liver disease(Child-Pugh C)
* Unstable angina and acute myocardium infarction
* Left ventricular ejection volume less than 30%,heart rate less than 50 beats per minute
* II and III degree atrioventricular block
* Systolic pressure less than 90 mmHg after giving vasopressors twice before beginning of this study
* Consciousness disturbance patients whose blood pressure less than 70mmHg and blood lactate more than 4.0mmol/L
* Suspected or confirmed long term use of narcotic analgesics
* Subjects who are breastfeeding or pregnant
* Allergic to investigational products or with other contraindication
* Participated in other study within 30 days

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-06 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Changes in blood pressure within 48 hours after drug intervention | Within 48 hours after drug intervention
Number of Participants with blood pressure decrease more than 20% of the baseline value or systolic pressure less than 100 mmHg | within 48 hours afer drug intervention
The number of cases who develop delirium | Within 48 hours after drug intervention

SECONDARY OUTCOMES:
Changes in heart rate | Within 48 hours after drug intervention
Changes in respiratory rate | Within 48 hours after drug intervention
Changes in central venous pressure | Within 48 hours after drug intervention